CLINICAL TRIAL: NCT02247011
Title: A 5-Year Long-term Follow-up Study of a Cross-Sectional Cohort Study (PK-VF) For the Examination of the Association of Vitamin D/Bone Turnover/Bone Mineral Density With an Incident Fracture in Chinese Postmenopausal Women
Brief Title: A 5-Year Follow-up Study Investigating Factors Associated With Osteoporotic Fracture in Chinese Postmenopausal Women
Acronym: PK-VF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: XWB-MISP-PKVF
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Osteoporotic Fractures; Osteoporosis, Postmenopausal
Keywords: bone mineral density; 25(OH)D
MeSH Terms: conditions — Osteoporotic Fractures; Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fracture group (Other): Fracture group included participants with new fractures during the 5 year follow-up visit. Fracture consists of non-vertebral fracture and vertebral fracture, which were investigated by questionnaire survey and lateral radiographs, respectively.
  Interventions: Other: Questionaire survey; Radiation: Bone mineral density examination; Radiation: Vertebral fracture assessment; Other: Biochemical markers analysis
- non-fracture group (Other): Fracture group included participants without new fractures during the 5 year follow-up visit. Fracture consists of vertebral fracture and non-vertebral fracture, which were investigated by questionnaire survey and lateral radiographs, respectively.
  Interventions: Other: Questionaire survey; Radiation: Bone mineral density examination; Radiation: Vertebral fracture assessment; Other: Biochemical markers analysis

INTERVENTIONS:
Other: Questionaire survey — We used a questionnaireto collect clinical data of the subjects. The questionnaire includes basic data, menstruation and pregnancy, habits and customs, daily activity, common healthy situation, history of drugs and history of factures.
Radiation: Bone mineral density examination — We use dual energy X-ray absorptiometry (DXA) to exam the BMD at lumbar spine (L2-4, LS) and hip.
Radiation: Vertebral fracture assessment — X-ray of thoracic and lumbar spine was taken, and the pictures were read by radiological specialists. The diagnosis of vertebral fracture was executed according to Genant's semiquantitative technique.
Other: Biochemical markers analysis — Fasting blood sample was collected for each subject. Common biochemical maerkers including serum calcium(Ca), serum phosphate(P), serum glucose(Glu), serum creatinine(Cr), alkaline phosphatase(ALP), alanine aminotransferase(ALT) were analyzed. Besides, we also detect bone speficific markers including 25-hydroxyl Vitamin D(25OHD), parathyroid hormone(PTH), β-isomerized C-terminal telopeptide of type I collagen(β-CTX), N-terminal procollagen of type 1 collagen(P1NP) and osteocalcin(OC).

SUMMARY:
This proposed study was designed to investigate the prevalence of a 5-year incident osteoporotic fracture and evaluate the association of a 5-year change of 25-hydroxyvitamin D (25[OH]D)/bone turnover makers/bone mineral density (BMD) with the incident fracture in the Chinese postmenopausal women, based on an endeavor of a 5-year post-baseline follow-up visit of a previous cross-sectional study, PK-VF, in which 1724 participants were enrolled and examined.

DETAILED DESCRIPTION:
1. In 2013, 5 years after PK-VF, the same 2070 subjects were contacted by the original sites. Among them 1242 subjects were able to come for the follow-up assessment.
2. Clinical assessments: The participant's bio-information, physical examination and medical history were collected;Questionnaire including social/life style and medical evaluations (years since menopause (YSM), fracture history, milk/yoghourt/coffee/wine intake, calcium intake, or smoking history) were collected by PK-VF investigators. Non-vertebral fracture history evaluation: specific non-vertebral fracture sites include rib or clavicle, forearm, upper arm, hand (including wrist), pelvis, hip, thigh (not including hip), leg, and foot (including ankle). When non-vertebral fractures are suspected, questions were raised to the participant to eliminate possible biases (How did you get these fractures, a slight fall at home, fell from a high place, hit by someone, broken during a car accident or an operation? Did you see a doctor to confirm these fractures?) A fracture occurred in regular daily activities or due to mild trauma was defined as fragile non-vertebral fracture.
3. Biochemical measurements: Fasting blood sample (~5 ml) was collected from each participant at participating sites; In 2007-2008 study, blood samples were collected during April-July, while in the 5-year follow-up; samples were collected in the same period of time. C-terminal telopeptide of type I collagen (β-CTX), N-aminoterminal prepeptide of type I procollagen (P1NP), and 25 (OH) D will be determined by a laboratory method of electrochemiluminescence (E170; Roche Diagnostics, Basel, Switzerland) in the institute (Peking Union); Chemistry including alkaline phosphatase (ALP), calcium (Ca), creatinine (Cr), and glucose, will be measured by using automated techniques in the institute (Peking Union);
4. BMD measurements: Lumbar spine (LS) and femoral neck (FN) BMDs by dual-energy x-ray absorptiometry (DXA) (Lunar or Norland) at PK-VF sites. BMD calibration: The participant's BMD were evaluated by the same type of DXA as previous. The coefficients of variation of the seven hospitals were 0.75% to 1.7% for LS and 0.56% to 1.0% for FN. Cross-calibration equations between machines are: LS BMD (g/cm^2) Lunar = 1.012 × Norland + 0.0137 and, FN BMD (g/cm^2) Lunar = 1.0377 × Norland + 0.00026
5. Vertebral fracture diagnosis: Lateral radiographs of the thoracolumbar spine (T4-L5) were taken at PK-VF sites. Vertebral fractures will be assessed using Genant's semi-quantitative visual criteria. Two specialist radiologists will independently evaluate and diagnose vertebral fracture. A worsened existing vertebral fracture will be regarded as a new vertebral fracture.

In 2007-2008 study(Published article about this study could be found in Pubmed, PMID: 24760246), 2070 participants were recruited in this cohort, and 837 subjects (40%) were diagnosed as osteoporosis. After 5 years, 1242 subjects agreed to be re-evaluated in 2013. Questionnaires and blood samples were collected, and BMD and spine x-ray were obtained at the 5-year follow up. We estimate that around 625 subjects would be diagnosed as osteoporosis. The remaining works include blood sample test (25(OH)D, CTX and P1NP),spine x-ray films reading, data input and statistical analysis, paper writing and publication.

ELIGIBILITY:
Inclusion Criteria:

1. postmenopausal women (normally over 50 years old and years since menopause over than 1 year) in Peking.
2. participants without any fracture in 2007 PK-VF study were included in the prospective study investigating the association of bone turnover markers/BMD/25(OH)D with fracture incidence.

Exclusion Criteria: participants with years since menopause less than 1 year.

Ages: 50 Years to 108 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weibo Xia, MD, Study Chair — Department of Endocrinology, Peking Union Medical College Hospital
Locations (1):
- Department of Endocrinology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In 2007-2008, 2070 postmenopausal women participated in the previous PK-VF study. After 5 years, 1100 subjects agreed to be re-evaluated in 2013.
Pre-assignment Details: All participants who agreed to be re-evaluated were enrolled in this study.
Groups:
- Overall Subjects: In 2007-2008, 2070 postmenopausal women participated in the previous PK-VF study. After 5 years, 1100 subjects agreed to be re-evaluated in 2013. Questionnaires and blood samples were collected, and BMD and spine x-ray were obtained from these 1100 participants.
Period: Overall Study
Arm/Group | Overall Subjects
Started | 1100
Completed | 975
Not Completed | 125
Not completed — Poor quality of radiological results | 125

BASELINE CHARACTERISTICS:
Groups:
- Non-fracture Group: Non-fracture group included participants without new fractures during the 5 year follow-up visit. Fracture consists of vertebral fracture and non-vertebral fracture, which were investigated by questionnaire survey and lateral radiographs, respectively.
- Total: Total of all reporting groups
Arm/Group | Fracture Group | Non-fracture Group | Total
Number analyzed (Participants) | 111 | 864 | 975
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70.08 [64.23 to 76.81] | 66.09 [59.84 to 74.59] | 66.72 [60.09 to 74.66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 864 | 975
  Male | 0 | 0 | 0
Years since menopause [Median (Inter-Quartile Range); unit: years] | 21.36 [12.87 to 29.59] | 16.43 [9.52 to 24.9] | 16.92 [9.98 to 25.28]
Previous osteoporotic fracture [Number; unit: participants]
  Previous osteoporotic fracture | 72 | 288 | 360
  No previous osteoporotic fracture | 39 | 576 | 615
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 25.21 (5.04) | 25.47 (4.85) | 25.46 (4.82)

OUTCOME MEASURES:

1. Primary Outcome: Non-vertebral Fracture Incidence
Description: Non-vertebral fractures were assessed by questionnaire survey.The overall incidence of non-vertebral fracture of the subjects is 7.18%( 70/975).
Time Frame: 5 year
Population: In 1100 participants, 975 of them finished the questionnaire
Measure: Number; unit: participants
Arm/Group | Fracture Group | Non-fracture Group
Number analyzed (Participants) | 111 | 864
participants | 70 | 0

2. Primary Outcome: Vertebral Fracture Incidence
Description: Vertebral fractures were assessed by lateral radiograph. The overall incidence of vertebral fracture of the subjects is 5.23%( 51/975)
Time Frame: 5 year
Measure: Number; unit: participants
Arm/Group | Fracture Group | Non-fracture Group
Number analyzed (Participants) | 111 | 864
participants | 51 | 0

3. Primary Outcome: Bone Mineral Density
Description: bone mineral density of Lumbar spine and femoral neck were measured by dual-energy X-ray absorptiometry (DXA) (Lunar or Norland)
Time Frame: 5 year
Measure: Median (Inter-Quartile Range); unit: g/cm^2
Arm/Group | Fracture Group | Non-fracture Group
Number analyzed (Participants) | 111 | 864
g/cm^2
  Lumbar spine BMD | 0.907 [0.784 to 1.015] | 0.956 [0.837 to 1.086]
  Femoral neck BMD | 0.686 [0.611 to 0.755] | 0.732 [0.647 to 0.820]
  Total hip BMD | 0.788 [0.736 to 0.845] | 0.845 [0.760 to 0.936]

4. Primary Outcome: Bone Turnover Markers and 25(OH)D
Description: C-terminal telopeptide of type I collagen (β-CTX), N-aminoterminal prepeptide of type I procollagen (P1NP), and 25-hydroxyvitamin D (25[OH]D) will be determined by a laboratory method of electrochemiluminescence (E170; Roche Diagnostics, Basel, Switzerland) in the institute (Peking Union)
Time Frame: 5 year
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Fracture Group | Non-fracture Group
Number analyzed (Participants) | 111 | 864
ng/ml
  β-CTX | 0.437 [0.309 to 0.529] | 0.401 [0.285 to 0.540]
  P1NP | 51.88 [41.40 to 70.16] | 51.57 [39.76 to 67.82]
  25(OH)D | 13.21 [10.00 to 17.43] | 12.49 [9.25 to 16.31]

5. Primary Outcome: Biochemical Markers
Description: Fasting blood sample was collected for each subject. Common biochemical markers including serum calcium(Ca), serum phosphate(P), serum glucose(Glu), serum creatinine(Cr), alkaline phosphatase(ALP)were analyzed.
Time Frame: 5 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fracture Group | Non-fracture Group
Number analyzed (Participants) | 111 | 864
mmol/L
  Serum calcium | 2.302 (0.565) | 2.263 (0.625)
  Serum phosphate | 1.148 (0.220) | 1.122 (0.345)
  Serum glucose | 6.083 (1.810) | 6.112 (1.281)

6. Primary Outcome: Serum Alkaline Phosphatase
Description: Fasting blood sample was collected for each subject. The level of serum alkaline phosphatase (ALP) was analyzed.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fracture Group | Non-fracture Group
Number analyzed (Participants) | 111 | 864
U/L | 79.4 (33.0) | 77.5 (37.0)

7. Primary Outcome: Serum Creatinine
Description: Fasting blood sample was collected for each subject.The level of serum creatinine(Cr) was analyzed.
Time Frame: 5 years
Measure: Mean (Standard Error); unit: umol/l
Arm/Group | Fracture Group | Non-fracture Group
Number analyzed (Participants) | 111 | 864
umol/l | 62.77 (17.73) | 64.91 (14.59)

ADVERSE EVENTS:
Groups:
- Overall Subjects: In 2007-2008, 2070 postmenopausal women participated in the previous PK-VF study. After 5 years, 1100 subjects agreed to be re-evaluated in 2013. Questionnaires and blood samples were collected, and BMD and spine x-ray were obtained from these 1100 participants. Of all these participants, 975 participants finished the questionnaire and for 961 of them, the spine x-ray was of enough quality to determine if there is vertebral fracture.
Arm/Group | Overall Subjects
Serious Adverse Events (participants affected / at risk) | 0/975
Other Adverse Events (participants affected / at risk) | 0/975

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes